CLINICAL TRIAL: NCT05994625
Title: Economic Evaluation of Stream™ Platform for the Early Detection of Anastomotic Leakage After Gastrointestinal Surgery
Brief Title: Economic Evaluation of Stream™ Platform
Acronym: CostAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FluidAI Medical (Industry)
Collaborators: Hamilton Health Sciences Corporation (Other); Ontario Bioscience Innovation Organization (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLS0007
Record Dates: First submitted 2023-07-18; First posted 2023-08-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Stream™ Platform will be attached to the abdominal/pelvic drains of the patients enrolled in this group. The platform will conduct continuous pH and electrical conductivity measurements of the abdominal drain fluid. The continuous pH and electrical conductivity measurements will be used to calculate a Risk Score that will be provided to surgeons. Surgeons will employ the Risk Score produced alongside the standard of care for guiding the postoperative care of patients.
  Interventions: Device: Stream™ Platform
- Control Group (Sham Comparator): Stream™ Platform will be attached to the abdominal/pelvic drains of the patients enrolled in this group. The platform will conduct continuous pH and electrical conductivity measurements of the abdominal drain fluid. However, Stream™ Platform will not generate a Risk Score and therefore, will not impact the postoperative care of patients. All procedures will be conducted as per the standard of care or institutional policies. Stream™ Platform will only be used for observation in the Control group.
  Interventions: Device: Stream™ Platform with Risk Score Omitted

INTERVENTIONS:
Device: Stream™ Platform — Stream™ Platform consists of 3 main components: Origin™ , Delta™ Monitor, and Stream™ Application. Origin™ is an inline biosensor system that can be attached inline between an off-the-shelf drainage catheter and reservoir system and is designed to monitor real-time changes in drained effluent characteristics (specifically pH and electrical conductivity (EC)) to identify potential anastomotic leaks. The Stream™ Application is a mobile application for displaying and analyzing data collected continuously via Origin™. Stream™ Application is pre-installed on Android mobile devices (called Delta™ Monitor).
  Stream™ Platform utilizes the continuous measurements of drain effluent characteristics to generate a Risk Score that is provided to the surgeon. The Risk Score is intended to provide an additional tool for the early diagnosis of anastomotic leakage.
  Arms: Intervention Group
Device: Stream™ Platform with Risk Score Omitted — Stream™ Platform consists of 3 main components: Origin™ , Delta™ Monitor, and Stream™ Application. Origin™ is an inline biosensor system that can be attached inline between an off-the-shelf drainage catheter and reservoir system and is designed to monitor real-time changes in drained effluent characteristics (specifically pH and electrical conductivity (EC)) to identify potential anastomotic leaks. The Stream™ Application is a mobile application for displaying and analyzing data collected continuously via Origin™. Stream™ Application is pre-installed on Android mobile devices (called Delta™ Monitor).
  This version of Stream™ Platform is utilized purely for observational purposes. Therefore, no Risk Score is generated. This allows postoperative monitoring of patients without any influence from the Stream™ Platform.
  Other Names: NERv's Inline Device
  Arms: Control Group

SUMMARY:
This Economic Evaluation study is a multi-center, two-arm, non-randomized, interventional trial. The purpose of this study is to evaluate the economic and patient outcomes of using the Stream™ Platform for early detection of anastomotic leakage after gastrointestinal surgery. The trial will track patient outcomes and healthcare costs in two groups: the intervention group, where the Stream platform is deployed, and the control group, before the integration of the Stream™ Platform. The data collected from both groups will be compared to assess the impact of implementing the Stream™ Platform and early leak detection on overall patient outcomes and healthcare costs.This trial will include hepatobiliary, colorectal, and trauma/acute care patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - Male or Female
* Subject understands and has voluntarily signed and dated the informed consent form (ICF).
* Subjects must be willing to comply with trial requirements
* Subject has performed an open or laparoscopic surgery with peritoneal or pelvic drainage

Exclusion Criteria:

* Subject is pregnant
* Subject will be discharged < 8 hours post-surgery
* 24 or more have passed since the end of the subject's surgery
* Involvement in the planning and conduct of the clinical investigation
* Subject is allergic to contrast medium
* Participation in another investigational drug or device study which would interfere with the endpoints of this study
* Device does not attach to drain used on the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Does Stream™ Platform integrate well with the existing clinical workflow (1)? | Through study completion, an average of 1 year
  Quantify average time spent by clinical research coordinator (CRC)/delegate interacting with Stream™ Platform (during attachment, daily calibration, and detachment) in minutes
Does Stream™ Platform integrate well with the existing clinical workflow (2)? | Through study completion, an average of 1 year
  Observe overall compliance to Instructions for use though quantification of the number of daily calibrations completed
Does Stream™ Platform integrate well with the existing clinical workflow (3)? | Through study completion, an average of 1 year
  Quantify the overall reported satisfaction score of the CRC/delegate through surveys.
Does Stream™ Platform reduce the cost of care for anastomotic leak patients in colorectal, hepatobiliary, and trauma and acute care surgeries (1)? | Upon study completion (12 months)
  Quantify the average number of tests and procedures performed to detect anastomotic leakage before and after the implementation of Stream™ Platform.
Does Stream™ Platform reduce the cost of care for anastomotic leak patients in colorectal, hepatobiliary, and trauma and acute care surgeries (2)? | Upon study completion (12 months)
  Quantify the average patient cost/cost of hospitalization and by-department cost (log of all billed items including medications, laboratory investigations, diagnostic/radiology investigations, hospital length of stay, ICU admission, re-admission within 30 days after discharge, time of discharge and therapeutic services) for colorectal, HPB, and trauma and acute care patients before and after the implementation of Stream™ Platform.
Number of Subjects with Device Related Adverse Events | Upon study completion (12 months)
  An adverse event assessment will be performed in accordance to ISO 14155 standards to determine the number of device related adverse events.

SECONDARY OUTCOMES:
Does Stream™ Platform allow for earlier postoperative anastomotic leak detection in colorectal, HPB, and trauma and acute care surgeries compared to clinical judgment/laboratory assessment (1)? | Upon study completion (12 months)
  Quantify the average time to detect anastomotic leakage after colorectal, HPB, and trauma and acute care patients using conventional diagnostic techniques (PRE) and after the implementation of Stream™ Platform (POST).
Does Stream™ Platform allow for earlier postoperative anastomotic leak detection in colorectal, HPB, and trauma and acute care surgeries compared to clinical judgment/laboratory assessment (2)? | Upon study completion (12 months)
  Quantify the average sensitivity, specificity, and overall accuracy of conventional diagnostic techniques for detection of anastomotic leakage after colorectal, HPB, and trauma and acute care surgeries in contrast to the average sensitivity, specificity, and overall accuracy of Stream™ Platform.
Does Stream™ Platform reduce the need for non-conservative management and hospital re-admission that is associated with anastomotic leak patients in colorectal, HPB, and trauma and acute care surgeries (1)? | Upon study completion (12 months)
  a. Quantify the average rate of type of re-intervention due to anastomotic leakage after colorectal, HPB, and trauma and acute care surgeries before and after the implementation of Stream™ Platform.
Does Stream™ Platform reduce the need for non-conservative management and hospital re-admission that is associated with anastomotic leak patients in colorectal, HPB, and trauma and acute care surgeries (2)? | Upon study completion (12 months)
  Quantify the average number of emergency re-admissions within 30 days after discharge due to anastomotic leakage in colorectal, HPB, and trauma and acute care surgeries before and after the implementation of Stream™ Platform.
Does Stream™ Platform reduce adverse events that are associated with anastomotic leak patients in colorectal, HPB, and trauma and acute care surgeries? | Upon study completion (12 months)
  Quantify the average number of adverse events (such as rate of secondary postoperative complications, rate of permanent stoma, 30-day mortality, etc.) due to anastomotic leakage after leakage in colorectal, HPB, and trauma and acute care surgeries before and after the implementation of Stream™ Platform.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Hamilton General Hospital - Hamilton Health Sciences, Hamilton, Ontario
  - Juravinski Hospital- Hamilton Health Sciences, Hamilton, Ontrario

IPD SHARING:
Plan to Share IPD: No